CLINICAL TRIAL: NCT05476809
Title: A Clinical Trial on an Upgraded Smart Cloth Home Care System With Interactive Family Caregiver App for Persons With Dementia
Brief Title: Upgraded Smart Cloth Home Care System for Persons With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 111-2314-B-182 -010 -MY3
Record Dates: First submitted 2022-07-26; First posted 2022-07-27 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-10

CONDITIONS: Dementia; Family
Keywords: dementia; family caregiver; smart care; home nursing
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: Current study plan to developed an advanced version of this smart-clothes care model based on prior study and the theory of Finding a Balance Point to further include monitoring for medication, abnormal life patter of the persons with dementia, and quality of hired care, and an interactive family caregiver app, and to examine this upgraded smart-clothes care system in a clinical trial.
Who Masked: Participant, Outcomes Assessor
Masking Description: Randomization to groups will follow a randomization table created by our university statistician. The project manager will create sequentially numbered sealed envelopes containing group assignment. Each consenting patient and their family caregiver will receive the envelope in the order in which they are enrolled. The project manager will have access to the spreadsheet that indicates the randomization order, but not the research nurses who assess outcomes. After randomization, patients and their family caregivers in the experimental group will receive the SCM, and those in the control group will receive usual care. Patients and families will not be aware of their group enrollment and will be masked to the care model they receive. Research nurses who collect data will be independent of those who deliver the interventions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- smart-cloth (Experimental): The upgraded smart-cloth assisted home nursing integrate smart-cloth monitoring system, home nursing, and family caregiver feedback app. The persons living with dementia will be asked to wear a smart cloth 24 hours a day and will be monitored on abnormal activity level, going out alone, abnormal number of getting-up at night, fall risks. In addition, monitoring for medication, abnormal life pattern, quality of hired help will also be included. The warning signals, along with weekly summary and related information will be sent to the family caregiver interactive App after the assessment of the home care nurses to provide guidance for family care.
  Interventions: Behavioral: smart-cloth assisted home nursing
- usual care (No Intervention): Routine clinical care will be provided to the participants.

INTERVENTIONS:
Behavioral: smart-cloth assisted home nursing — The upgraded smart-cloth assisted home nursing integrate smart-cloth monitoring system, home nursing, and family caregiver feedback app. The persons living with dementia will be asked to wear a smart cloth 24 hours a day and will be monitored on abnormal activity level, going out alone, abnormal number of getting-up at night, fall risks. In addition, monitoring for medication, abnormal life pattern, quality of hired help will also be included. The warning signals, along with weekly summary and related information will be sent to the family caregiver interactive App after the assessment of the home care nurses to provide guidance for family care.
  Arms: smart-cloth

SUMMARY:
The purposes of this study are to develop an upgraded version of the smart-clothes home care model that include an interactive family caregiver App, and to examine its effect on a randomized controlled trial.

DETAILED DESCRIPTION:
The purposes of this study are to develop an upgraded version of the smart-clothes home care model that include an interactive family caregiver App, and to examine its effect on a randomized controlled trial. This 3-year study will spend the first 6 months to developed the upgraded smart-clothes home care model, and the later 2 and a half years on the clinical trial and follow-ups. In addition to the original function of abnormal activity level, going out alone, abnormal number of getting-up at night, fall risks, this upgraded version will include monitoring for medication, abnormal life pattern, quality of hired help. The warning signals, along with weekly summary and related information will be sent to the family caregiver interactive App after the assessment of the home care nurses to provide guidance for family care.

During the first 6 months, the upgraded smart-clothes home care model will be developed according to qualitative and quantitative data of the prior study and expert reviews. For the clinical trial in later 2 1/2 years, a total of 60 participant families will be randomly assigned to experimental (N=30) and control (N=30) group, with experimental group receiving the upgraded smart-clothes home care for 6 months and control group received routine care with 6 month follow-ups. Outcomes including caregiver preparedness, balance between competing needs, health related quality of life and depressive symptoms, and fall, time up & go, activities of daily living (ADLs), instrumental ADLs, cognitive function and quality of life of the patient will be followed every 2 month for 6 months. Intention-to-treat and hierarchical linear models will be used to analyze the results.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as having dementia
* can walk independently or with help
* able to communicate
* living in Northern Taiwan.
* Family caregiver age 20 or older
* taking primary responsibility in providing family care.

Exclusion Criteria:

* with terminal illness
* with severe diseases that can not be controlled.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
caregiver preparedness | baseline
  Preparedness is measured by self-report with an 8-item scale. This scale asks caregivers to rate how well-prepared they think they are for seven domains of caregiving.
caregiver preparedness | 2 months after baseline
  Preparedness is measured by self-report with an 8-item scale. This scale asks caregivers to rate how well-prepared they think they are for seven domains of caregiving.
caregiver preparedness | 4 months after baseline
  Preparedness is measured by self-report with an 8-item scale. This scale asks caregivers to rate how well-prepared they think they are for seven domains of caregiving.
caregiver preparedness | 6 months after baseline
  Preparedness is measured by self-report with an 8-item scale. This scale asks caregivers to rate how well-prepared they think they are for seven domains of caregiving.
caregiver depressive symptoms | baseline
  Centre for Epidemiologic Studies Depression Scale (CES-D)
caregiver depressive symptoms | 2 months after baseline
  Centre for Epidemiologic Studies Depression Scale (CES-D)
caregiver depressive symptoms | 4 months after baseline
  Centre for Epidemiologic Studies Depression Scale (CES-D)
caregiver depressive symptoms | 6 months after baseline
  Centre for Epidemiologic Studies Depression Scale (CES-D)
Caregiving Balance | Baseline
  The degree of balance between competing needs will be measured by the Caregiving Process of Finding a Balance Point measure (Shyu, 2002).
Caregiving Balance | 2 month after Baseline
  The degree of balance between competing needs will be measured by the Caregiving Process of Finding a Balance Point measure (Shyu, 2002).
Caregiving Balance | 4 month after Baseline
  The degree of balance between competing needs will be measured by the Caregiving Process of Finding a Balance Point measure (Shyu, 2002).
Caregiving Balance | 6 month after Baseline
  The degree of balance between competing needs will be measured by the Caregiving Process of Finding a Balance Point measure (Shyu, 2002).
Caregiving Health Related Quality of Life | Baseline
  Medical Outcome SF-36 Taiwan version
Caregiving Health Related Quality of Life | 2 month after Baseline
  Medical Outcome SF-36 Taiwan version
Caregiving Health Related Quality of Life | 4 month after Baseline
  Medical Outcome SF-36 Taiwan version
Caregiving Health Related Quality of Life | 6 month after Baseline
  Medical Outcome SF-36 Taiwan version

SECONDARY OUTCOMES:
Time Up and Go test | baseline
  assessing fall risk for the persons living with dementia
Time Up and Go test | 2 month after baseline
  assessing fall risk for the persons living with dementia
Time Up and Go test | 4 month after baseline
  assessing fall risk for the persons living with dementia
Time Up and Go test | 6 month after baseline
  assessing fall risk for the persons living with dementia (PLWD)
Activities of Daily Living (ADL) | baseline
  Chinese Barthel Index leasing independence in ADL for PLWD
Activities of Daily Living (ADL) | 2 months after baseline
  Chinese Barthel Index leasing independence in ADL for PLWD
Activities of Daily Living (ADL) | 4 months after baseline
  Chinese Barthel Index leasing independence in ADL for PLWD
Activities of Daily Living (ADL) | 6 months after baseline
  Chinese Barthel Index leasing independence in ADL for PLWD
Instrumental activities of daily living (IADL) | baseline
  Lawton and Brody's IADL measure
Instrumental activities of daily living (IADL) | 2 months after baseline
  Lawton and Brody's IADL measure
Instrumental activities of daily living (IADL) | 4 months after baseline
  Lawton and Brody's IADL measure
Instrumental activities of daily living (IADL) | 6 months after baseline
  Lawton and Brody's IADL measure
Cognitive function | baseline
  Mini-Mental State Examination
Cognitive function | 2 month after baseline
  Mini-Mental State Examination
Cognitive function | 4 month after baseline
  Mini-Mental State Examination
Cognitive function | 6 month after baseline
  Mini-Mental State Examination
Health related quality of life for PLWD | baseline
  Medical Outcomes SF-36 Taiwan Version
Health related quality of life for PLWD | 2 month after baseline
  Medical Outcomes SF-36 Taiwan Version
Health related quality of life for PLWD | 4 month after baseline
  Medical Outcomes SF-36 Taiwan Version
Health related quality of life for PLWD | 6 month after baseline
  Medical Outcomes SF-36 Taiwan Version

CONTACTS AND LOCATIONS:
Overall Officials: Yea-Ing L Shyu, PhD, Principal Investigator — Professor
Locations (2):
- Taiwan (2):
  - New Taipei Tucheng hospital, New Taipei City
  - Chang Gung Memorial Hospital, Taiwan, Taoyuan District

IPD SHARING:
Plan to Share IPD: No